CLINICAL TRIAL: NCT00605748
Title: PV-Isolation for Paroxysmal Atrial Fibrillation: Isolation of the Arrhythmogenic Vein(s) vs. Isolation of All Veins
Brief Title: Pulmonary Vein (PV) -Isolation: Arrhythmogenic Vein(s) Versus All Veins
Acronym: PAVAV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Prof. A. Schömig, Deutsches Herzzentrum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GE IDE No. C00807
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Last update posted 2008-08-27 (Estimated); Status verified 2008-08

CONDITIONS: Atrial Fibrillation
Keywords: catheter ablation; atrial fibrillation; pulmonary vein
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Segmental PV-Isolation of the arrhythmogenic vein(s)
  Interventions: Procedure: Segmental PV-Isolation of the arrhythmogenic vein(s)
- 2 (Active Comparator): Segmental PV-Isolation of all veins
  Interventions: Procedure: Segmental PV-Isolation of all veins

INTERVENTIONS:
Procedure: Segmental PV-Isolation of the arrhythmogenic vein(s) — isolation of pulmonary veins for curing atrial fibrillation
  Arms: 1
Procedure: Segmental PV-Isolation of all veins — isolation of pulmonary veins for curing atrial fibrillation
  Arms: 2

SUMMARY:
We conduct a randomized study comparing the safety and effectiveness of two interventional ablation techniques for treatment of paroxysmal atrial fibrillation: the segmental pulmonary vein ablation approach, (1) with empiric isolation of all pulmonary veins or (2) Segmental Isolation of the arrhythmogenic pulmonary vein(s)

DETAILED DESCRIPTION:
BACKGROUND Atrial fibrillation ablation procedures typically involve isolation of all pulmonary veins (PVs), yet the need for such an extensive ablation strategy in all patients is unclear.

OBJECTIVE:

We conduct a randomized study comparing the safety and effectiveness of two interventional ablation techniques for treatment of paroxysmal atrial fibrillation: the segmental pulmonary vein ablation approach, (1) with empiric isolation of all pulmonary veins or (2) Segmental Isolation of only the arrhythmogenic pulmonary vein(s). The single-blind interventional, randomized study will include 106 patients in each arm.

A reablation procedure, with the use of the same technique as the first ablation, will be offered to the patient in case of a symptomatic atrial fibrillation recurrence beyond the third month after the ablation procedure.

Follow-Up After discharge, patients w ill be scheduled for repeated visits in the arrhythmia clinic at 3 and 6 months after the first ablation. At each of these visits, intensive questioning for arrhythmia-related symptoms (fatigue, dizziness, and nausea) since the last follow-up visit was performed, especially for those that the patient had experienced before ablation. At every follow-up visit, 7-day Holter monitoring w ill be performed. Multislice CT or MRI of the pulmonary vein w ill be obtained before and 3 months after the ablation procedure for evaluation of the pulmonary vein anatomy and for detection of radiofrequency ablation-induced pulmonary vein stenosis .

Study End Points and Definitions The primary end point of the study will be freedom from atrial tachyarrhythmias (of > 30-second duration) including atrial fibrillation and atypical atrial flutter documented by 7-day Holter monitoring performed at the 6-month follow-up. Two secondary study end points will be chosen. The first will be freedom from arrhythmia-related symptoms during the 6-month follow-up. Because early recurrences of atrial tachyarrhythmias within the first month after ablation may be a transient phenomenon, this time interval was excluded from analysis. Second, a composite of periprocedural pericardial tamponade, thromboembolic complications, and pulmonary vein stenosis with > 50% lumen loss (main vessel or first branching) was defined as a safety end point

ELIGIBILITY:
Inclusion Criteria:

* patients between 18 and 80 years old with paroxysmal atrial fibrillation
* Episodes with a maximum duration for 7 days
* at least 4 episodes / month
* at least one attempt with Class I or III anti-arrhythmic drugs and/or with ß-blockers without success
* sufficient oral anticoagulation for a minimum of four weeks previous to ablation

Exclusion Criteria:

* hyperthyroidism
* mitral regurgitation > II°
* intracardiac thrombi documented by transesophageal echocardiography
* left ventricular ejection< fraction 35%,
* history of ablation, myocardial infarction or cardiac surgery in the previous 3 months
* history of left-atrial ablation procedure
* contraindication for oral anticoagulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
freedom of atrial tachycardia 6 months after ablation | 6 months

SECONDARY OUTCOMES:
freedom of symptoms due to atrial tachycardia 6 months after ablation safety | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Deisenhofer, MD, Study Chair — Deutsches Herzzentrum Muenchen; Heidi L. Estner, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Germany

REFERENCES:
- [Derived] Fichtner S, Hessling G, Ammar S, Reents T, Estner HL, Jilek C, Kathan S, Buchner M, Dillier R, Deisenhofer I. A prospective randomized study comparing isolation of the arrhythmogenic vein versus all veins in paroxysmal atrial fibrillation. Clin Cardiol. 2013 Jul;36(7):422-6. doi: 10.1002/clc.22132. Epub 2013 May 13. PMID 23670880